CLINICAL TRIAL: NCT00673114
Title: A Prospective, Phase I/II Trial Determining the Efficacy and Safety of Allogeneic Hematopoietic Stem Cell Transplantation Using Banked Unrelated Umbilical Cord Blood Supplemented With Related, Haplo-Identical T-Cell Depleted Stem Cells in Subjects With High Risk Malignancies
Brief Title: Unrelated Cord Blood Transplant Plus a Haplo-Identical (Half-Matched), T-Cell Depleted Stem Transplant From a Related Donor for Subjects With High Risk Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008292; 8717 (Other: Duke Legacy IRB Number)
Record Dates: First submitted 2007-12-27; First posted 2008-05-07 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Hematologic Malignancy; Myelodysplastic Syndrome (MDS); Aplastic Anemia
Keywords: Haplo/cord; hematologic malignancy; MDS; Aplastic Anemia; AML; ALL; CML
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant Recipients (Other)
  Interventions: Biological: haplo/cord transplant

INTERVENTIONS:
Biological: haplo/cord transplant — T-cell depleted haplo-matched cells from related donor and unrelated umbilical cord blood

SUMMARY:
Subjects will be diagnosed with a hematological malignancy (cancer of the blood), which is unlikely to be cured with conventional non-transplant therapy. The best results of bone marrow transplant are obtained with the donor is a relative that has identical tissue type (HLA-type). These subjects will not have such a donor available but they will have a appropriately matching unrelated umbilical cord blood unit (UCB). However, the cord blood unit does not contain a high enough number of cells and may take longer to engraft (or grow). The purpose of this study is to determine whether the addition of stem cells from a family member to supplement a standard unrelated cord blood transplant is safe and will increase the success of the cord blood transplantation procedure. Subjects enrolled in this study will receive an unrelated cord blood transplant plus a haplo-identical (half-matched), T-cell depleted stem transplant from a related donor. The goal of this study is to determine whether the addition of the related stem cells accelerates bone marrow recovery and improves long-term disease free survival.

DETAILED DESCRIPTION:
Over the past decade, umbilical cord blood transplantation has been shown to be a viable alternative donor stem cell source for hematopoietic cell transplantation in subjects with catastrophic diseases treatable with transplantation therapy. UCB cells can cross partially mismatched HLA barriers without intolerable acute or chronic Graft-versus-Host Disease(GVHD). Thus, many subjects lacking a sufficiently matched, living related or unrelated bone marrow or adult stem cell donor, can use partially HLA-matched UCB cells for stem cell rescue after myeloablative irradiation and/or chemotherapy. UCB Cell dose, expressed per kilogram of recipient body weight, is the best predictor of outcomes after UCB transplantation. Cell dose thresholds strongly correlating with outcomes have been identified.

In subjects receiving lower cell doses, while durable engraftment will ultimately occur, there are significant delays in myeloid and platelet engraftment which, at best, result in longer hospitalization and significant increases in resource utilization and in the worst cases, result in increased early deaths from infection and regimen-related toxicity.

In infants and children weighing <40kg, it is possible to find a sufficiently matched UCB unit that will deliver a dose of cells critical for successful engraftment (defined as 5 x 10^7 nucleated cells/kg) within a reasonable time frame in >90% of subjects. In teenagers and adults weighing >40kg, this is not always possible. Because UCB units contain a relatively fixed number of total nucleated cells, units delivering optimal cell dosing for subjects weighing >70kg will only be identified <10% of the time. Attempts to increase the dose of cells available for UCBT have included ex vivo expansion and combined unit transplantation. While expansion of UCB cells ex vivo is possible, infusion of these expanded cells have not resulted in shortening of engraftment times. Likewise, combinations of up to 5 UCB units for a single myeloablative transplant have not shortened time to neutrophil or platelet engraftment.

In this study, we take an alternative approach to facilitating early myeloid engraftment in subjects undergoing UCB transplantation therapy. In subjects who cannot only identify a donor delivering a cell dose >2 x 10^7 nucleated cells/kg, we will augment the UCBT with a lower dose of haplo-identical, T-cell depleted stem cells from a related adult donor to facilitate early, short-term engraftment with the primary goal of minimizing early infections and other non-relapse mortality while the UCB cells engraft as the durable and permanent graft. As the immunocompetent UCB cells engraft, we expect that they will reject the immunologically incompetent haplo-identical adult stem cells. Thus, after approximately 100-180 days post transplant, the subject should convert to 100% donor chimerism with the UCB donor graft.

In this study, we will investigate the use of unrelated UCB obtained from the umbilical cord blood banks supplements with related, haplo-identical, T-cell depleted stem cells in subjects with high risk refractory malignancies, myelodysplasia or severe aplastic anemia amenable to stem cell transplantation therapy but lacking conventional related or unrelated donors.

OBJECTIVES:

1. To determine the safety of co-transplantation of unrelated umbilical cord blood supplemented with related, haplo-identical, T-cell depleted stem cells in subjects with high risk malignancies.
2. To describe the rates of neutrophil and platelet engraftment and immune reconstitution in these subjects.
3. To determine whether short and long term lymphohematopoietic engraftment is derived from one or both donor sources.

The primary endpoint of the study is number of days to ANC of 500/uL

The secondary endpoints of the study are:

1. 180 day survival
2. Non-relapse mortality in the first 180 days post transplant
3. Number of days to untransfused platelet count of 50K/uL
4. Incidence of primary and secondary graft failure
5. Incidence and severity of acute and chronic graft-versus-host disease (GVHD)
6. Pace and quality of immune reconstitution
7. Rates of leukemic relapse
8. Donor chimerism

ELIGIBILITY:
Inclusion Criteria:

* Patient Selection Criteria: Patients with high risk or refractory malignancies, myelodysplasia (MDS) or severe aplastic anemia amenable to stem cell transplantation therapy but lacking conventional related or unrelated donors will be eligible for this trial.
* Have a consenting related haplo-identical (3/6 or 4/6) stem cell donor;
* Have an available 3, 4, 5, or 6/6 antigen matching unrelated UCB unit that will deliver a cell dose between 2.0-5.0 x 10e7cells/kg.
* Not have a consenting 6/6 or 5/6 antigen matched related bone marrow donor or genetically matched unrelated BM or adult stem cell donor.
* Patients must be <55 years of age at the time of study enrollment.
* Patients must have histologically confirmed diagnosis of a hematologic malignancy, MDS or severe aplastic anemia. Eligible patients include the following:
* Patients with high risk ALL in first complete remission, with high risk being defined by the presence of hypodiploidy, t(4;11; MLL. 11q23) or t(9;22), or patients presenting with extreme hyperleukocytosis (initial WBC >500,000/ml) or failure to achieve a complete remission after standard induction therapy.
* All patients with ALL or ANLL in second or subsequent remission.
* Patients with ALL or ANLL in relapse.
* Patients with MDS.
* Patients with CML in any chronic phase, accelerated phase or blast crisis.
* Patients with severe aplastic anemia refractory to medical therapy.
* Patients must not have active CNS disease at the time of study enrollment.
* Patients must have a good performance status (Lansky 80-100%, Karnofsky 50-100%).
* Patients must have adequate function of other organ systems as measured by:
* Creatinine < 2.0 mg/dl and creatinine clearance > 50 cc/min/m2.
* Hepatic transaminases (ALT/AST) < 4 x normal, bilirubin < 2.0 mg/dl.
* Normal cardiac function by echocardiogram or radionuclide scan, (ejection fraction or shortening fraction > 80% of normal value for age).
* Pulmonary function tests demonstrating FVC and FEV1 of >60% of predicted for age. For adult patients DLCO > 60% of predicted. If patient cannot perform PFTs, clearance by the pediatric or adult pulmonologist will be required.
* Patients must not have uncontrolled infections at the time of cytoreduction.
* Patient, parent, or legal guardian must have given written informed consent according to FDA guidelines.
* Patients may not be pregnant or lactating and must have a current negative pregnancy test.
* Patients must have a minimum life expectancy of at least 3 months.
* Patients must have an available related haplo-identical stem cell donor and an available unrelated cord blood donor delivering between 2 x10e7 cells/kg and 5 x 10e7 cells/kg and matching at a minimum of 3/6 HLA loci.
* Patients must be HIV negative.
* Patients must not be concurrently involved in any other clinical trial that affects engraftment or immune reconstitution (e.g. other hematopoietic growth factors).
* Patients must not have any co-morbid condition which, in the view of the Principal Investigators, renders the patient at too high a risk from treatment complications and regimen related morbidity/mortality.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2007-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University Medical Center Pediatric Blood and Marrow Transplant
Locations (1):
- Duke University Medical Center Pediatric Blood and Marrow Transplant, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three patients enrolled.
Groups:
- Transplant Recipients: Transplant Recipients
Period: Overall Study
Arm/Group | Transplant Recipients
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Transplant Recipients: single arm study
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Reaching Primary Endpoint of Absolute Neutrophil Count (ANC) of 500/uL (Engraftment).
Time Frame: By day 100
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
participants | 3

2. Secondary Outcome: 180 Day Survival
Description: Number of participants alive at 180 days post transplant
Time Frame: 180 days
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
participants | 3

3. Secondary Outcome: Non-Relapse Mortality at 180 Days Post Transplant
Time Frame: 180 days
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
participants | 0

4. Secondary Outcome: Platelet Engraftment (Untransfused and Platelet Count > 50,000)
Description: Participants platelet engrafted.
Time Frame: Approximately 1 year
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
participants | 3

5. Secondary Outcome: Incidence of Primary and Secondary Graft Failure
Description: Number of participants experiencing graft failure.
Time Frame: 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
participants | 0

6. Secondary Outcome: Number of Participants With Acute or Chronic Graft-versus-host Disease (GVHD)
Description: Acute and chronic GVHD
Time Frame: two years
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
participants | 2

7. Secondary Outcome: Rates of Leukemic Relapse
Description: Number of participants relapsed
Time Frame: Up to 2 years post transplant
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
participants | 1

8. Secondary Outcome: Number of Participants With Donor Cells at 100 Days Post-transplant
Time Frame: Post transplant
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Arm/Group | Transplant Recipients
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Recipients (N=3)
Encephalitis infection (Infections and infestations) | 1 (1) — Not study related and not unexpected per the PI.
Chronic GVHD (General disorders) | 1 (1) — Not directly related to the study and not unexpected per the PI.
Relapse (Blood and lymphatic system disorders) | 1 (1) — Not study related and not unexpected per the PI.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not directly related to the study and not unexpected per the PI.
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not directly related to the study and not unexpected per the PI.
Multi-system organ failure (General disorders) | 1 (1) — Not directly related to the study and not unexpected per the PI.
Sepsis (Infections and infestations) | 1 (1) — Not directly related to the study and not unexpected per the PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes